CLINICAL TRIAL: NCT02560155
Title: Preoperative Decolonization and Surgical Site Infections - a Prospective Randomized Trial (DECO-SSI Trial)
Brief Title: Preoperative Decolonization and Surgical Site Infections - a Prospective Randomized Trial
Acronym: DECO-SSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenhofgruppe AG (Industry)
Collaborators: Clinical Trials Unit Bern (CTU) (Unknown); Lindenhofstiftung (Unknown); Labormedizinisches Zentrum Dr. Risch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-11-F
Record Dates: First submitted 2015-09-16; First posted 2015-09-25 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Orthopedic Disorders; Surgical Site Infection
Keywords: Orthopedic surgery; Surgical site infection; Decolonization; Staphylococcus aureus
MeSH Terms: conditions — Musculoskeletal Diseases; Surgical Wound Infection; Staphylococcal Infections | interventions — Mupirocin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nose-SA-carriers control (No Intervention): Control Group, no intervention
- Nose-SA-carriers decolonized (Active Comparator): Chlorhexidine sol 4%; Mupirocin 2% nasal ointement
  1 shower/day for 5 days and Nasal ointement 2x/d in each nostril for 5 days preoperatively
  Interventions: Drug: Mupirocin 2% nasal ointement; Drug: Chlorhexidine sol 4%
- Non-nose-SA-carriers control (No Intervention): Control Group, no intervention
- Non-nose-carriers decolonized (Active Comparator): Chlorhexidine sol 4% shower, daily for 5 days preoperatively
  Interventions: Drug: Chlorhexidine sol 4%

INTERVENTIONS:
Drug: Mupirocin 2% nasal ointement — Mupirocin nasal ointement 2x/d for 5 days preoperatively
  Other Names: Bactroban Nasal
  Arms: Nose-SA-carriers decolonized
Drug: Chlorhexidine sol 4% — Shower with Chlorhexidine sol 4% once a day for 5 days preoperatively
  Other Names: Lifo-Scrub sol 4%
  Arms: Non-nose-carriers decolonized; Nose-SA-carriers decolonized

SUMMARY:
Surgical site infections are a major postoperative complication and are mostly due to colonization with endogenous germs, like Staphylococcus aureus, Staphylococcus epidermidis or Propionibacterium acnes. In literature, preoperative decolonization procedures showed a trend in lowering surgical site infection rates, but especially in orthopedic surgery data is controversial and randomized controlled trials are lacking. In the main study, the study investigators aim at performing a controlled prospective randomized interventional trial to measure the impact of preoperative decolonization of nasal Staphylococcus aureus carriers on surgical site infection rates in orthopedic surgery. In an alongside study a controlled prospective randomized interventional trial to measure the impact of preoperative skin decolonization of patients undergoing an orthopedic procedure will be conducted.

DETAILED DESCRIPTION:
All participants will be assessed for eligibility during preoperative othopedic consultation. 2-3 weeks prior operation date participants will be screened for Staph. aureus carriage by nose-swab. According to nose-swab results randomizaton and allocation to study arm will be performed.

After one and three months post-operatively participants will be asked by phone interview if surgical site infections occured. Results have to be confirmed by orthopedic surgeon if possible.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 16 years
* patient undergoing elective orthopedic procedure at the Sonnenhof hospital
* decolozination protocol can be performed timely
* signed informed consent

Exclusion Criteria:

* no orthopedic surgery planned
* allergy to mupirocin or chlorhexidine
* presence of a nasal foreign body
* no informed consent
* pregnancy
* decolozination protocol can't be followed timely
* patients undergoing treatment/surgery for a documented infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Overall number of participants with surgical site infections 3 months postoperatively | 3 months
  Phone interview and orthopedic assessement

SECONDARY OUTCOMES:
Number of participants with surgical site infections at 1 and 3 months postoperatively | 1 and 3 months
  Phone interview and orthopedic assessement

OTHER OUTCOMES:
Total screening costs | one year
  Total screening costs divided by the number of prevented SSI to assess cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brügger, Dr. med., Principal Investigator — Lindenhofgruppe AG
Locations (1):
- Sonnenhofspital, Lindenhofgruppe, Bern, Switzerland